CLINICAL TRIAL: NCT00519025
Title: Risk Factors for Linezolid Resistance in Staphylococcus Aureus
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Brian Potoski, Assistant Professor, University of Pittsburgh
Other Study IDs: PRO07080006; investigator funding (Other: UPMC)
Record Dates: First submitted 2007-08-17; First posted 2007-08-21 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Linezolid Resistance; Staphylococcus Aureus
Keywords: Linezolid; Staphylococcus Aureus; Infections
MeSH Terms: conditions — Staphylococcal Infections; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a retrospective chart review study. The proposed study aims to document the risk factors for quinolone resistance in bloodstream isolates of Klebsiella species. Additionally, the adequacy of empiric antibiotic therapy for Klebsiella bloodstream infections will be assessed.

DETAILED DESCRIPTION:
This is a retrospective chart review study. The proposed study aims to document the risk factors for quinolone resistance in bloodstream isolates of Klebsiella species. Additionally, the adequacy of empiric antibiotic therapy for Klebsiella bloodstream infections will be assessed. This research is important because identification of risk factors may allow earlier initiation of appropriate therapy in patients infected with these bacteria. Additionally, we will identify whether horizontal spread is responsible for this increasing trend.

ELIGIBILITY:
Inclusion Criteria:

* patients with linezolid resistance to staphylococcus aureus

Exclusion Criteria:

* those that don't meet entry criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: linezolid resistance to staph aureus
Sampling Method: Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2007-08 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Potoski, PharmD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States